CLINICAL TRIAL: NCT00739817
Title: Screening for Primary Ciliary Dyskinesia Using Nasal Nitric Oxide
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Israel Amirav, Ziv Medical center
Other Study IDs: HP-6-199-R
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background: Primary ciliary dyskinesia (PCD) is a rare genetic disease characterised by recurrent respiratory infections and subfertility due to dysfunction of cilia (brushes) of the lining cells. Undiagnosed and untreated it can result in an irreversible crippling chronic lung disease. The diagnosis of PCD is a difficult one and involves the complex assessment of ciliary structure and function. Thus, PCD is under diagnosed and appropriate preventative and symptomatic treatment may be denied in many patients. In addition, the gene responsible for PCD is at present unknown, thus preventing pre-natal diagnosis and genetic counseling.

Working hypothesis and aims: Recently, it has become apparent that the evaluation of nasally expired nitric oxide (NO) constitutes a simple and non-invasive diagnostic method, which discriminates between PCD patients, PCD carriers and healthy controls at high rate of specificity and sensitivity. Testing is simple and last approximately one minute. We have recently identified a unique isolated Druze population with high prevalence of PCD. The high frequency of disease places this closed community at a high risk of undiagnosed PCD.

The aim of this project is to use nasal NO measurement as a screening tool to identify possible undiagnosed cases of PCD and PCD carriers in this high risk Druze population.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary willing to participate

Exclusion Criteria:

* Recent URTI
* Steroids use 2 weeks prior to testing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2010-07

PRIMARY OUTCOMES:
Nasal NO < 105 ppb | at enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Department, Ziv Medical Center, Safed, Israel